CLINICAL TRIAL: NCT01671852
Title: A Randomized Controlled Trial of Intranasal Mometasone in Children With Obstructive Sleep Apnea Due to Adenotonsillar Hypertrophy
Brief Title: Intranasal Mometasone in Children With Obstructive Sleep Apnea Due to Adenotonsillar Hypertrophy
Acronym: Nasonex OSA
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Could not obtain funding.
Sponsor: Children's & Women's Health Centre of British Columbia (Other)
Responsible Party: Principal Investigator, Neil Chadha, Dr. Neil K. Chadha MBChB(Hons),MPHe BSc(Hons),FRCS, Children's & Women's Health Centre of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H12-01653
Record Dates: First submitted 2012-07-05; First posted 2012-08-24 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Obstructive Sleep Apnea (Mild, Moderate, Severe) as Per Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Lymphoma, Follicular | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasonex (Active Comparator): The intervention group will receive mometasone nasal sprays at the dosage outlined below for 8 weeks. For patients that are between age 3 to 11 years and if they are randomized to the medicated group, they will use pediatric dosing of Mometasone nasal sprays, 1 spray (50 mcg) in each nostril once daily for 8 weeks. For patients that are older than age 12 and if they are randomized to the medicated group, they will use adult dosing of Mometasone nasal sprays, 2 sprays (100mcg) in each nostril twice daily for 8 weeks.
  Interventions: Drug: Mometasone furoate nasal spray
- Saline (Placebo Comparator): The placebo group will receive saline nasal sprays for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone furoate nasal spray — Included patients will be randomized to a sequence of treatments including a medicated nasal spray and a saline nasal spray. The medicated group will receive Mometasone nasal sprays at the dosage outlined below for 8 weeks. The placebo group will receive saline nasal sprays for an equal duration. Informed consent of the parents or legal guardians will be obtained.
  For patients that are between age 3 to 11 years and if they are randomized to the medicated group, they will use pediatric dosing of Mometasone nasal sprays, 1 spray (50 mcg) in each nostril once daily for 8 weeks. For patients that are older than age 12 and if they are randomized to the medicated group, they will use adult dosing of Mometasone nasal sprays, 2 sprays (100mcg) in each nostril twice daily for 8 weeks.
  Other Names: Nasonex
  Arms: Nasonex
Drug: Placebo
  Arms: Saline

SUMMARY:
Obstructive sleep apnea (OSA) in children is a disorder of breathing during sleep characterized by prolonged partial upper airway obstruction and/or intermittent complete obstruction (obstructive apnea) that disrupts normal breathing during sleep1. The condition occurs in 2-5% of children and can occur at any age, but it is most common in children between the ages of 2 to 62,3. Untreated OSA is associated with lung disease, heart disease, growth delay, poor learning and behavioral problems such as inattention and hyperactivity. The most common underlying risk factor for the development of OSA is enlargement of tonsils and adenoids. Given the potential risk of complications associated with surgery of the tonsils and adenoids, medications to shrink the adenoids without requiring surgery have been considered, in particular intranasal corticosteroids (INCSs) which is a nose spray. A recent Cochrane systematic review suggested a short-term benefit of INCSs in children with mild to moderate OSA4. The authors recommended that further randomised controlled studies were required to evaluate the efficacy of INCSs in children with OSA. In particular they recommended that future studies should employ sleep studies to look for any improvement with INCSs, and should include children with more severe OSA, as these are the patients at the greatest risk of complications of surgery and would benefit most from a non-surgical treatment. The purpose of this study is therefore to explore the efficacy of INCSs in children with the full spectrum of OSA severity, including sleep study analysis., and longer term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children between age 3 and 16 with objectively diagnosed OSA (mild, moderate, severe) as per polysomnography (AHI ≥ 1/h, where AHI is the sum of obstructive and mixed apneas and obstructive hypopneas).

Exclusion Criteria:

* Children with malformation syndromes or craniofacial anomalies
* Children with neuromuscular disorders
* Children with morbid obesity (body mass index ≥ 40)
* Children with asthma requiring steroid treatment

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | 8 weeks
  This wil be measured by polysomnography.

SECONDARY OUTCOMES:
Respiratory Disturbance Index | At baseline and after each phase of treatment (i.e. after initial 8 weeks invention and again after second 8 weeks intervention)
  This will be measured by polysomnography.
Desaturation index | At baseline and after each phase of treatment (i.e. after initial 8 weeks invention and again after second 8 weeks intervention)
  This will be measured by polysomnography.
Respiratory arousal index | At baseline and after each phase of treatment (i.e. after initial 8 weeks invention and again after second 8 weeks intervention)
  This will be measured by polysomnography.
Nadir of arterial oxygen saturation | At baseline and after each phase of treatment (i.e. after initial 8 weeks invention and again after second 8 weeks intervention)
  This will be measured by polysomnography.
Mean arterial oxygen saturation | At baseline and after each phase of treatment (i.e. after initial 8 weeks invention and again after second 8 weeks intervention)
  This will be measured by polysomnography.
Avoidance of surgical treatment for OSA | At baseline and after each phase of treatment (i.e. after initial 8 weeks invention and again after second 8 weeks intervention)
  This will be measured by polysomnography.
Clinical symptom score (based on parent repot of, for example, snoring, witnessed apnea, daytime sleepiness etc.) | At baseline and after each phase of treatment (i.e. after initial 8 weeks invention and again after second 8 weeks intervention)
  This will be measured by polysomnography.
Tonsillar size (on an ordinal scale from 0 [not visible] to +4 [tonsils touch]) | At baseline and after each phase of treatment (i.e. after initial 8 weeks invention and again after second 8 weeks intervention)
  This will be measured by polysomnography.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Women's and Children's Hospital, Vancouver, British Columbia, Canada